CLINICAL TRIAL: NCT05006677
Title: Effectiveness and Safety of Different Antithrombotic Therapy for the Treatment of Ventricular Thrombus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-TR
Record Dates: First submitted 2021-08-08; First posted 2021-08-16 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Ventricular Thrombus
MeSH Terms: interventions — acarboxyprothrombin; Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-vitamin K antagonist oral anticoagulants (NOACs)
  Interventions: Drug: non-vitamin K antagonist oral anticoagulants (NOACs)
- vitamin K antagonists (VKAs)
  Interventions: Drug: vitamin K antagonists (VKAs)
- antiplatelet agents
  Interventions: Drug: antiplatelet agents
- non-antithrombotic therapy
  Interventions: Other: non-antithrombotic therapy

INTERVENTIONS:
Drug: non-vitamin K antagonist oral anticoagulants (NOACs) — Collecting information of patients with VT who received NOACs
  Groups: non-vitamin K antagonist oral anticoagulants (NOACs)
Drug: vitamin K antagonists (VKAs) — Collecting information of patients with VT who received VKAs
  Groups: vitamin K antagonists (VKAs)
Drug: antiplatelet agents — Collecting information of patients with VT who received antiplatelet agents
  Groups: antiplatelet agents
Other: non-antithrombotic therapy — Collecting information of patients with VT without any antithrombotic therapy
  Groups: non-antithrombotic therapy

SUMMARY:
To observe the effectiveness and safety of different therapies-non-vitamin K antagonist oral anticoagulants (NOACs) or vitamin K antagonists (VKAs) or antiplatelet agents and non-antithrombotic therapy - for the treatment of VT.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ventricular thrombus(VT), regardless of sex, basic diseases, occupation or education;
* The VT should be found newly within 3 months;
* The observational phase should last until the time that patients who had achieved thrombus resolution. The following up period after the phase ended should continue for at least 3 months.

Exclusion Criteria:

* Individuals received standard antithrombotic therapy within 4 weeks;
* Individuals received the thrombectomy therapy, ventricular aneurysm resection or heart transplantation within 6 weeks since the VT was found in the first time;
* Had a long history of VT more than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a diagnosis of VT in Fuwai Hospital, National Center of Cardiovascular Diseases in China from July 2010 through March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Thrombus resolution in 12 weeks follow-up | 12 weeks
  Thrombus resolution in 12 weeks follow-up

SECONDARY OUTCOMES:
Thrombus resolution in 6 weeks follow-up | 6 weeks
  Thrombus resolution in 6 weeks follow-up
Thrombus resolution in 6 months follow-up | 6 months
  Thrombus resolution in 6 months follow-up
Thrombus resolution in 12 months follow-up | 12 months
  Thrombus resolution in 12 months follow-up
Thromboembolism events | 12 months
  Thromboembolism events
Bleeding | 12 months
  Bleeding
All-cause death | 12 months
  All-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Qing Yang, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gianstefani S, Douiri A, Delithanasis I, Rogers T, Sen A, Kalra S, Charangwa L, Reiken J, Monaghan M, MacCarthy P. Incidence and predictors of early left ventricular thrombus after ST-elevation myocardial infarction in the contemporary era of primary percutaneous coronary intervention. Am J Cardiol. 2014 Apr 1;113(7):1111-6. doi: 10.1016/j.amjcard.2013.12.015. Epub 2014 Jan 14. PMID 24485697
- [Background] Turpie AG, Robinson JG, Doyle DJ, Mulji AS, Mishkel GJ, Sealey BJ, Cairns JA, Skingley L, Hirsh J, Gent M. Comparison of high-dose with low-dose subcutaneous heparin to prevent left ventricular mural thrombosis in patients with acute transmural anterior myocardial infarction. N Engl J Med. 1989 Feb 9;320(6):352-7. doi: 10.1056/NEJM198902093200604. PMID 2643772
- [Background] Abdelnaby M, Almaghraby A, Abdelkarim O, Saleh Y, Hammad B, Badran H. The role of rivaroxaban in left ventricular thrombi. Anatol J Cardiol. 2019 Jan;21(1):47-50. doi: 10.14744/AnatolJCardiol.2018.48313. No abstract available. PMID 30587707
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] He J, Ge H, Dong JX, Zhang W, Kong LC, Qiao ZQ, Zheng Y, Ding S, Wan F, Shen L, Wang W, Gu ZC, Yang F, Li Z, Pu J. Rationale and design of a prospective multi-center randomized trial of EARLY treatment by rivaroxaban versus warfarin in ST-segment elevation MYOcardial infarction with Left Ventricular Thrombus (EARLY-MYO-LVT trial). Ann Transl Med. 2020 Mar;8(6):392. doi: 10.21037/atm.2020.02.117. PMID 32355836
- [Background] Guddeti RR, Anwar M, Walters RW, Apala D, Pajjuru V, Kousa O, Gujjula NR, Alla VM. Treatment of Left Ventricular Thrombus With Direct Oral Anticoagulants: A Retrospective Observational Study. Am J Med. 2020 Dec;133(12):1488-1491. doi: 10.1016/j.amjmed.2020.05.025. Epub 2020 Jun 27. PMID 32598904
- [Derived] Yang Q, Liang Y, Quan X, Lang X, Gao D. Characteristics of Novel Anticoagulants versus Vitamin K Antagonists in the Ventricular Mural Thrombus. Rev Cardiovasc Med. 2023 Mar 2;24(3):74. doi: 10.31083/j.rcm2403074. eCollection 2023 Mar. PMID 39077494
- [Derived] Yang Q, Quan X, Lang X, Liang Y. Predicting Thromboembolism in Hospitalized Patients with Ventricular Thrombus. Rev Cardiovasc Med. 2022 Nov 30;23(12):390. doi: 10.31083/j.rcm2312390. eCollection 2022 Dec. PMID 39076670
- [Derived] Yang Q, Lang X, Quan X, Gong Z, Liang Y. Different Oral Antithrombotic Therapy for the Treatment of Ventricular Thrombus: An Observational Study from 2010 to 2019. Int J Clin Pract. 2022 Feb 24;2022:7400860. doi: 10.1155/2022/7400860. eCollection 2022. PMID 35685496